CLINICAL TRIAL: NCT01075516
Title: TARIFF Health Economics Evaluation Registry for Remote Follow up
Brief Title: Health Economic Evaluation of Remote Follow up for Implantable Cardioverter Defibrillator (ICD) Patients
Acronym: TARIFF
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR 09 021 IT RC
Record Dates: First submitted 2010-02-02; First posted 2010-02-25 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Complication of Cardiac Defibrillator
Keywords: Remote Monitoring; ICD patients; EQ-5D questionnaire; remote follow up

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard Follow Up: ICD patients followed through periodic in-hospital visits
- Remote Follow Up: ICD patients followed with remote transmitters (Merlin@Home) that periodically communicate correct system functioning

SUMMARY:
The purpose of the study is to define the economic value of implantable cardioverter defibrillator (ICD) remote monitoring for hospitals, third payers and patients in Italy. Aims of the study are to develop a hospital cost minimization analysis and a cost effectiveness analysis based on direct estimation of costs and quality of life deriving from remote follow-up (performed with Merlin@home and Merlin.net) compared to standard follow-up in the management of ICD implanted patients.

DETAILED DESCRIPTION:
TARIFF is a prospective observational study aimed to measure direct, indirect costs and quality of life of all participants for the duration of the observational timeframe. Purpose of cost collecting is to include a complete set of medical services and productivity loses that could be directly affected by the different clinical Follow-Up (FU) pathway. The study consists of 2 phases: firstly standard follow up costs will be collected for 100 pts, then all costs associated to remote follow ups will be collected for other 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients already implanted with ICD
* Patients able to be followed in the same centre during all the study
* Patients with age > 18
* Patients able to understand and to answer to EuroQoL Group 5-Dimension (EQ-5D) Questionnaire

Exclusion Criteria:

* Patients pregnant
* Patients unable to connect Merlin@home transmitters with Website Merlin.net (i.e.without telephonic analogic line or Global System for Mobile Communication (GSM)/Universal Mode Telecommunication System (UMTS) connection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with ICD according to current guidelines and with the possibility to use Merlin@home transmitters
Sampling Method: Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Santini, Prof., Principal Investigator — Ospedale San Filippo Neri, Roma, Italy
Locations (6):
- Italy (6):
  - Azienda Ospedaliera S.Gerardo, Monza, Monza (MB)
  - Casa di Cura Pederzoli, Peschiera del Garda, VR
  - Ospedale Careggi, Florence
  - Ospedale Luigi Sacco, Milan
  - Ospedale Monaldi, Napoli
  - Ospedale San Filippo Neri, Roma

REFERENCES:
- [Background] Wilkoff BL, Auricchio A, Brugada J, Cowie M, Ellenbogen KA, Gillis AM, Hayes DL, Howlett JG, Kautzner J, Love CJ, Morgan JM, Priori SG, Reynolds DW, Schoenfeld MH, Vardas PE; Heart Rhythm Society; European Heart Rhythm Association; American College of Cardiology; American Heart Association; European Society of Cardiology; Heart Failure Association of ESC; Heart Failure Society of America. HRS/EHRA expert consensus on the monitoring of cardiovascular implantable electronic devices (CIEDs): description of techniques, indications, personnel, frequency and ethical considerations. Heart Rhythm. 2008 Jun;5(6):907-25. doi: 10.1016/j.hrthm.2008.04.013. No abstract available. PMID 18551743
- [Background] Morichelli L, Ricci RP. Remote monitoring of implantable devices: the European experience. Heart Rhythm. 2009 Jul;6(7):1077-80. doi: 10.1016/j.hrthm.2009.02.030. Epub 2009 Feb 24. No abstract available. PMID 19560096
- [Background] Ricci RP, Morichelli L, Santini M. Remote control of implanted devices through Home Monitoring technology improves detection and clinical management of atrial fibrillation. Europace. 2009 Jan;11(1):54-61. doi: 10.1093/europace/eun303. Epub 2008 Nov 16. PMID 19011260
- [Background] Marzegalli M, Lunati M, Landolina M, Perego GB, Ricci RP, Guenzati G, Schirru M, Belvito C, Brambilla R, Masella C, Di Stasi F, Valsecchi S, Santini M. Remote monitoring of CRT-ICD: the multicenter Italian CareLink evaluation--ease of use, acceptance, and organizational implications. Pacing Clin Electrophysiol. 2008 Oct;31(10):1259-64. doi: 10.1111/j.1540-8159.2008.01175.x. PMID 18811805
- [Background] Ricci RP, Morichelli L, Santini M. Home monitoring remote control of pacemaker and implantable cardioverter defibrillator patients in clinical practice: impact on medical management and health-care resource utilization. Europace. 2008 Feb;10(2):164-70. doi: 10.1093/europace/eum289. Epub 2008 Jan 16. PMID 18199570
- [Background] Seto E. Cost comparison between telemonitoring and usual care of heart failure: a systematic review. Telemed J E Health. 2008 Sep;14(7):679-86. doi: 10.1089/tmj.2007.0114. PMID 18817497
- [Background] Clark RA, Inglis SC, McAlister FA, Cleland JG, Stewart S. Telemonitoring or structured telephone support programmes for patients with chronic heart failure: systematic review and meta-analysis. BMJ. 2007 May 5;334(7600):942. doi: 10.1136/bmj.39156.536968.55. Epub 2007 Apr 10. PMID 17426062
- [Background] Lunati M, Gasparini M, Santini M, Landolina M, Perego GB, Pappone C, Marzegalli M, Argiolas C, Murthy A, Valsecchi S; InSync ICD Italian Registry Investigators. Follow-up of CRT-ICD: implications for the use of remote follow-up systems. Data from the InSync ICD Italian Registry. Pacing Clin Electrophysiol. 2008 Jan;31(1):38-46. doi: 10.1111/j.1540-8159.2007.00923.x. PMID 18181908
- [Background] Ricci RP, D'Onofrio A, Padeletti L, Sagone A, Vicentini A, Vincenti A, Morichelli L, Cavallaro C, Ricciardi G, Lombardi L, Fusco A, Rovaris G, Silvestri P, Guidotto T, Pollastrelli A, Santini M. Rationale and design of the health economics evaluation registry for remote follow-up: TARIFF. Europace. 2012 Nov;14(11):1661-5. doi: 10.1093/europace/eus093. Epub 2012 Apr 27. PMID 22544910
- [Result] Ricci RP, Vicentini A, D'Onofrio A, Sagone A, Vincenti A, Padeletti L, Morichelli L, Fusco A, Vecchione F, Lo Presti F, Denaro A, Pollastrelli A, Santini M. Impact of in-clinic follow-up visits in patients with implantable cardioverter defibrillators: demographic and socioeconomic analysis of the TARIFF study population. J Interv Card Electrophysiol. 2013 Nov;38(2):101-6. doi: 10.1007/s10840-013-9823-5. Epub 2013 Sep 21. PMID 24057266
- [Result] Ricci RP, Vicentini A, D'Onofrio A, Sagone A, Rovaris G, Padeletti L, Morichelli L, Fusco A, De Vivo S, Lombardi L, Denaro A, Pollastrelli A, Colangelo I, Santini M. Economic analysis of remote monitoring of cardiac implantable electronic devices: Results of the Health Economics Evaluation Registry for Remote Follow-up (TARIFF) study. Heart Rhythm. 2017 Jan;14(1):50-57. doi: 10.1016/j.hrthm.2016.09.008. Epub 2016 Sep 8. PMID 27614025

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The sample size defined at least 100 pts per arm. The protocol allows few patients over in each of the 2 arms.
Period: Overall Study
Arm/Group | Standard Follow Up | Remote Follow Up
Started | 107 | 102
Completed | 89 | 86
Not Completed | 18 | 16
Not completed — Death | 5 | 9
Not completed — Lost to Follow-up | 10 | 2
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Standard Follow-Up: Implantable cardioverter defibrillators (ICD) patients followed through periodic in-hospital visits
- Remote Follow-Up: ICD patients followed with remote transmitters (Merlin@Home) that periodically communicate correct system functioning
- Total: Total of all reporting groups
Arm/Group | Standard Follow-Up | Remote Follow-Up | Total
Number analyzed (Participants) | 107 | 102 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (11.5) | 69.7 (10.2) | 69.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 92 | 86 | 178
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — All Subjects enrolled in Italian centers. Number of subjects
  participants
    Italy | 107 | 102 | 209
Implant Indication [Count of Participants; unit: Participants]
  Primary Prevention | 83 | 82 | 165
  Secondary Precention | 24 | 20 | 44
New York Heart Association (NYHA) [Number; unit: participants] — Count of participants in each grade. "NYHA Functional Class provides a classification of heart failure based on symptomatic limitations to activities of daily living and ranges from NYHA Functional Class I to IV: NYHA Functional Class I is defined as no limitations in physical activity and NYHA Functional Class IV is defined as the presence of heart failure symptoms resulting in inability to carry out any physical activity without discomfort
  participants
    I | 25 | 30 | 55
    II | 51 | 33 | 84
    III | 28 | 38 | 66
    IV | 3 | 1 | 4
ejection fraction (EF)% [Mean (Standard Deviation); unit: percentage of blood] — EF% is an Echo derived measurements in percentage
  percentage of blood | 32.2 (10.6) | 31.8 (9.6) | 32.0 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Economic Impact of Remote Monitoring on Hospitals and Patients
Description: Costs analysis of remote monitoring using Merlin@home and Merlin.net compared to standard follow-up in an Italian real-life setting. Overall mean annual cost per patient: Health Care System (HCS) perspective.
Time Frame: 12 months follow-up
Measure: Mean (Standard Deviation); unit: Euro (€)
Arm/Group | Standard Follow Up | Remote Follow Up
Number analyzed (Participants) | 89 | 86
Euro (€) | 1044.89 (1990.47) | 482.87 (2488.10)
Statistical Analysis 1: Comparison: Standard Follow Up vs Remote Follow Up; Test type: Other — Continuous data summarized as mean ± Standard Deviation (SD). For cost data Wilcoxon rank-sum test was used to compare costs across groups. The analysis evaluated HCS perspective of group membership impact (SC vs RM) on total health care cost, adjusting for covariates that were significantly different between the groups at the .2 significance level. Differences between the 2 groups were assessed using differences in sample means (point estimates) and t distributions (confidence intervals); p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Impact of Remote Monitoring on Procedural Costs for the Italian Health Economic System (SSN)
Description: Comparison of Cardiovascular Hospitalizations costs for the Italian Health Economic System derived from the use of Merlin@Home system versus standard in clinic follow-up
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Euro (€)
Arm/Group | Standard Follow Up | Remote Follow Up
Number analyzed (Participants) | 89 | 86
Euro (€) | 886.67 (1979.13) | 432.34 (2487.86)
Statistical Analysis 1: Comparison: Standard Follow Up vs Remote Follow Up; Test type: Other — Continuous data are summarized as mean ± SD. For cost data the Wilcoxon rank-sum test was used to compare costs across groups. This analysis evaluated the impact of group membership (SC vs RM) on cardiovascular hospitalization timeframe (outcome), adjusting for covariates that were significantly different between the groups at the .2 significance level. Differences between the 2 groups were assessed using differences in sample means (point estimates) and t distributions (confidence intervals); p = 0.003, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Impact of Remote Monitoring on Patients' Quality of Life
Description: Evaluation of patient quality of life through Quality of Life (EQ-5D) questionnaire during follow up with/without using Merlin@Home system.
  Utility (patients' preferences) and Quality-adjusted life-year (QALY) scales were used. QALYs were based on utility, the EuroQoL EQ-5D-3L questionnaire was administered to each patient at baseline and at 12 months in order to calculate utility values (both ranges from 0 to 1). High score means better outcomes.
  One quality-adjusted life-year (QALY) is equal to 1 year of life in perfect health. QALYs are calculated by estimating the years of life remaining for a patient following a particular treatment or intervention and weighting each year with a quality-of-life score (on a 0 to 1 scale).
Time Frame: baseline, 12 months
Population: The clinical benefit for patients were evaluated through EQ-5D questionnaire. The results of the questionnaire were used to measure the quality-adjusted life years (QALY). It was considered costs and EQ-5D values only for the patients alive who completed the questionnaires (87 SC and 79 RM).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Follow Up | Remote Follow Up
Number analyzed (Participants) | 87 | 79
score on a scale
  Utility at baseline | 0.8621 (0.1853) | 0.8686 (0.1342)
  Utility at 12 months | 0.8463 (0.1846) | 0.8703 (0.1618)
  Quality Adjusted Life Years (Method 1) | 0.8542 (0.1689) | 0.8694 (0.1329)
Statistical Analysis 1: Comparison: Standard Follow Up vs Remote Follow Up; For the patient perspective, the quality of life associated with the 2 strategies was assessed. Quality of life is reported as utility values from the EuroQoL Group 5-Dimension 3-Level Self-Report (EQ-5D-3L) questionnaire and quality adjusted life years (QALYs) were based on utility (patients' preferences). The EQ-5D-3L questionnaire was administered to each patient at baseline and at 12 months in order to calculate utility values (from 0 to 1); Test type: Other — Continuous data are summarized as mean ± SD. This analysis evaluated the impact of group membership (SC vs RM) on total health care cost (outcome), adjusting for covariates that were significantly different between the groups at the .2 significance level. However, as the arithmetic mean is the most informative measurement for policy decisions, differences between the 2 groups were assessed using differences in sample means (point estimates) and t distributions (confidence intervals); p = 0.80, t-test, 2 sided — Comparison of utility at baseline from the EQ-5D-3L questionnaire
Statistical Analysis 2: Comparison: Standard Follow Up vs Remote Follow Up; For the patient perspective, the quality of life associated with the 2 strategies was assessed. Quality of life is reported as utility values from the EQ-5D-3L questionnaire and quality adjusted life years (QALYs) were based on utility (patients' preferences). The EQ-5D-3L questionnaire was administered to each patient at baseline and at 12 months in order to calculate utility values (from 0 to 1); Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.38, t-test, 2 sided — Comparison of utility at 12 months from the EQ-5D-3L questionnaire
Statistical Analysis 3: Comparison: Standard Follow Up vs Remote Follow Up; [analysis description as in outcome 3, analysis 2]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.53, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Standard Follow Up | Remote Follow Up
Serious Adverse Events (participants affected / at risk) | 21/107 | 34/102
Other Adverse Events (participants affected / at risk) | 18/107 | 18/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Follow Up (N=107) | Remote Follow Up (N=102)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 8 (10) | 3 (3)
Cardiac Death (General disorders) | 0 (0) | 3 (3)
Death (General disorders) | 2 (2) | 2 (2)
Unknown cause of death (General disorders) | 3 (3) | 4 (4)
Implant site infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pocket formation of decubitus (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Subdural Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Device inappropriate shock delivery (Product Issues) | 1 (1) | 3 (4)
Device stimulation issue (Product Issues) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 3 (3) | 6 (11)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 2 (2)
Cardioversion (Surgical and medical procedures) | 3 (3) | 2 (2)
Hospitalization (Surgical and medical procedures) | 2 (2) | 4 (5)
Medical device repositioning (Surgical and medical procedures) | 0 (0) | 1 (1)
Mitral Valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 3 (3) | 0 (0)
Syncope (Vascular disorders) | 0 (0) | 1 (1)
Cardiovascular event prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Motor disfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Colitis ulcerative (Immune system disorders) | 1 (1) | 0 (0)
Hemorrage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Follow Up (N=107) | Remote Follow Up (N=102)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 3 (3) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Eye symptoms (Eye disorders) | 2 (3) | 0 (0)
Blood pressure dicreased (Investigations) | 0 (0) | 1 (1)
Device capturing issue (Product Issues) | 0 (0) | 2 (2)
Device electrical impedence issue (Product Issues) | 0 (0) | 1 (1)
Device inappropriate shock delivery (Product Issues) | 3 (4) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 1 (1)
Device pacing issue (Product Issues) | 4 (6) | 5 (5)
Device stimulation issue (Product Issues) | 2 (4) | 2 (2)
Device telemetry issue (Product Issues) | 0 (0) | 5 (5)
Oversensing (Product Issues) | 2 (2) | 1 (1)
Undersensing (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No